CLINICAL TRIAL: NCT07046052
Title: A Double Blind Randomised Controlled Trial Comparing Continuous Infusion vs. Programmed Intermittent Bolus Via a Pericapsular Nerve Group (PENG) Catheter for Post Operative Fractured Neck of Femur Analgesia
Brief Title: PENG Block: Continuous Infusion vs. Programmed Intermittent Bolus in Neck of Femur Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Consultant Anaesthesiologist, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIB PENG RCT ECM5(3)5/3/2024
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hip Fracture; Analgesia Post Fracture
Keywords: hip fracture; regional anaesthesia; analgesia; peng block; continuous infusion; programmed intermittent bolus; randomised controlled trial
MeSH Terms: conditions — Hip Fractures; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous PENG Infusion (Active Comparator): Participants will be randomly assigned to this arm and will receive a continuous infusion of levobupivacaine.
  Interventions: Other: continuous infusion of levobupivacaine
- Programmed Intermittent Bolus PENG (Experimental): Participants will be randomly assigned to this arm and will receive a timed pre-set bolus dose of levobupivacaine.
  Interventions: Other: Programmed Intermittent Bolus of Levobupivacaine

INTERVENTIONS:
Other: continuous infusion of levobupivacaine — Participants in this arm will receive a continuous infusion of levobupivacaine via a regional anaesthesia catheter placed in the PENG fascial space. The total dose over 24 hours will be equivalent in both arms of the study.
  Arms: Continuous PENG Infusion
Other: Programmed Intermittent Bolus of Levobupivacaine — Participants in this arm will receive a timed pre-set bolus dose of levobupivacaine via a regional anaesthesia catheter placed in the PENG fascial space. The total dose over 24 hours will be equivalent in both groups.
  Arms: Programmed Intermittent Bolus PENG

SUMMARY:
Pericapsular Nerve Group Block (PENG) is an effective regional anaesthesia modality in providing analgesia following neck of femur fracture. Continuous PENG techniques, using indwelling catheters and infusions of local anaesthetic, facilitate the continuation of analgesia for a number of days following hip fracture surgery. It is unclear from the published literature whether an optimal strategy of local anaesthetic delivery has been characterized.

Similar doses of local anaesthetic agents can be administered by either continuous infusion or timed intermittent bolus. It is unclear whether one dosing strategy is superior to the other in the context of hip fracture analgesia. The study aims to evaluate the clinical efficacy of both dosing strategies in patients undergoing hip fracture surgery.

DETAILED DESCRIPTION:
The latest Irish Hip Fracture Database (IHFD) National Report published in 2020 counted 3,666 hip fractures in patients aged over 60 during the year 2020 across the Republic of Ireland. Ninety five percent of these patients received surgical fixation representing a significant clinical workload. Hip fractures are most often associated with increasing age and frailty and indeed 52% of patients included in the IHFD report were aged over 80 years. Fractures of the proximal femur are painful and, in the absence of regional analgesia, usually require strong opioids to control. Patients of this age group are more likely to suffer from cognitive impairment (31% in the IHFD cohort) and reduced renal function, both of which complicate opioid use making their avoidance desirable. Impaired renal function and ischaemic heart disease, which is also common in this cohort, also contraindicate non-steroidal anti-inflammatory drug (NSAID) use. Such limitations make analgesia challenging following hip fracture surgery and it is known that poor perioperative analgesia in this group increases the incidence of delirium, a factor independently associated with increased requirement for long term care and mortality. It is essential therefore that effective peri-operative analgesia is prioritised and provided in such a way that minimises potential cognitive, renal and cardiovascular complications. Regional analgesia provides a simple and effective way to ensure high-quality pain relief throughout the acute hip fracture journey whilst avoiding many of the complications associated with the use of systemic analgesia. Pre-operative ultrasound guided regional analgesia has now become the standard of care for patients presenting to the emergency department with fractured neck of femur. The recent procedure specific post operative pain management (PROSPECT) recommendations from the PROSPECT group and the European Society of Regional Anaesthesia and Pain Medicine (ESRA) regarding hip fracture repair surgery recommend either a single short femoral nerve block (FNB) or a fascia iliaca compartment block (FICB) due to their pain score lowering and opioid sparing effects2. They go on to say that there is currently insufficient evidence to recommend peri-capsular nerve group (PENG) blocks or the routine use of catheter-based techniques citing the potential for prolonged motor block being an additional concern for the latter. As such the PENG block and cathether-based techniques need to be studied in more detail to allow national and international guidance groups to make appropriate recommendations.

The nerve supply to the hip joint and surrounding structures is primarily via the femoral, obturator and accessory obturator nerves (L2 - L4) anteriorly and the sciatic nerve (L4 - S3) posteriorly. The superior and inferior gluteal nerves and the quadratus femoris nerve, branches of the sacral plexus, also contribute to the posterior innervation of the hip joint. The PENG block has been relatively recently described as a technique for analgesia following hip surgery as an alternative to more traditional regional analgesia techniques such as the FNB or FICB3. It involves placing local anaesthetic beneath the psoas tendon in the iliopsoas groove of the ilium and pubis bones between the anterior inferior iliac spine and the medial border of the iliopubic eminence. The aim of the block is to anaesthetise the articular branches of the obturator, accessory obturator and femoral nerves supplying the anterior capsule of the hip which run over or close to this groove and into the hip capsule3. These nerves are small and not easily visible on ultrasound and as such the end point of the block is local anaesthetic spread along the periosteal groove; for this reason the PENG block could be considered a fascial plane block. There is considerable anatomical variation between individuals in the number, origin, course and sensory supply of the articular branches of these nerves4, it is important therefore that relatively large volumes of local anaesthetic are used to ensure sufficient spread from the point of injection to reach the target nerves, indeed in the original description of the block the volume used was 20ml3. The PENG block theoretically has advantages over the FNB and FICB in that it only targets the articular branches and not the primary nerves and thus potentially has less effect on quadriceps power5,6. This has important implications for the early mobilisation and physiotherapy engagement post-operatively.

At our institution the current analgesic pathway for patients undergoing hemiarthroplasty surgery for fractured neck of femur includes a PENG block immediately before surgery. In almost all cases the patient also simultaneously receives a PENG catheter which is used into the post-operative period for ongoing regional analgesia. The infusion usually runs for approximately 48 - 72 hours with the patients being followed up daily by an acute pain team. All patients presenting to the hospital with fractured neck of femur also receive a single shot block, either a FNB or a FICB in the emergency department. This typically happens between 12 and 48 hours pre-operatively.

Programmed intermittent bolus (PIB) protocols involve the delivery of a set volume of local anaesthetic via a pump at a set time interval delivered as a bolus rather than a continuous infusion. There is strong evidence in the obstetric population for the benefits of programmed intermittent bolus (PIB) for labour epidural analgesia especially when combined with a patient controlled epidural analgesia (PCEA) element. Improved maternal satisfaction with analgesia as well as an overall reduction in total local anaesthetic infused are amongst the benefits which have led to many obstetric units switching over to the technique7 The evidence for PIB infusion techniques via peripheral nerve catheters is less well established however improved pain scores at 24 and 48 hours post operatively as well as improved patient satisfaction and decreased requirement for rescue analgesia have been reported8. The results are however conflicting, this is exacerbated by the wide gamut of different peripheral nerve blocks each with their own anatomical characteristics. It would seem logical that plane blocks, such as the PENG block, would benefit more from a PIB protocol given the importance of local anaesthetic spread in these techniques but this has also not been consistently shown7. There are promising results from studies of PIB vs. CI in thoracic paravertebral catheters (a block which similarly requires larger volumes of local anaesthetic for improved spread) for thoracic surgery9,10.

Previous literature reviews of intermittent bolus versus continuous infusions techniques have highlighted the paucity of evidence in this area and the heterogenicity of the patients and techniques in the few trials that are available7. Hip fracture represents an ideal index condition for studying this topic given the large numbers of patients and the frequent use of peripheral nerve catheters in this population. PENG catheters, being a relatively new technique, need to be assessed using a PIB protocol to establish its effectiveness in comparison to more traditional CI protocols. It is hoped that in conducting this trial we will be able to assess the efficacy of PIB techniques in PENG catheters used for analgesia following femoral hemiarthroplasty after fractured neck of femur.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* over the age of 18 years
* hemiarthroplasty for fractured neck of femur
* able to provide written consent.

Exclusion Criteria:

* under 50kg body weight.
* unable to provide consent due to incapacity
* pregnant women
* vulnerable adults under state guardianship
* Patients with pre-existing chronic pain disorders or with a history of long-term opioid use
* those with contraindications to a peripheral nerve block such as local site infection, allergy to local anaesthetic or those who are coagulopathic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Pain Scale (NRS 0-10) | 48 Hours Post-operatively
  Patients will be invited to rate their post operative pain at rest and on movement on a 0-10 scale; where 0 is no pain and 10 is worst imaginable pain.

SECONDARY OUTCOMES:
Numeric Rating Pain Scale (NRS 0-10) | 1, 2, 4, 24 hours postoperatively
Quality of Recovery 15 (QOR15) | 48 hours postoperatively
  Patients will be invited to complete a validated multidomain assessment of recovery following anaesthesia and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin P Atterton, MBChB FRCA, Study Director — Cork University Hospital & University College Cork
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
We have not considered making IPD available but would consider doing so with appropriate data security safeguards in place with collaborators on request.

REFERENCES:
- [Background] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023
- [Background] Lin X, Liu CW, Goh QY, Sim EY, Chan SKT, Lim ZW, Chan DXH. Pericapsular nerve group (PENG) block for early pain management of elderly patients with hip fracture: a single-center double-blind randomized controlled trial. Reg Anesth Pain Med. 2023 Nov;48(11):535-539. doi: 10.1136/rapm-2022-104117. Epub 2023 Apr 13. PMID 37055189
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Yang L, Huang X, Cui Y, Xiao Y, Zhao X, Xu J. Combined Programmed Intermittent Bolus Infusion With Continuous Infusion for the Thoracic Paravertebral Block in Patients Undergoing Thoracoscopic Surgery: A Prospective, Randomized, and Double-blinded Study. Clin J Pain. 2022 Jun 1;38(6):410-417. doi: 10.1097/AJP.0000000000001037. PMID 35442613
- [Background] Chen L, Wu Y, Cai Y, Ye Y, Li L, Xia Y, Papadimos TJ, Xu X, Wang Q. Comparison of programmed intermittent bolus infusion and continuous infusion for postoperative patient-controlled analgesia with thoracic paravertebral block catheter: a randomized, double-blind, controlled trial. Reg Anesth Pain Med. 2019 Feb;44(2):240-245. doi: 10.1136/rapm-2018-000031. Epub 2019 Jan 5. PMID 30700619
- [Background] Law WZW, Sara RA, Cameron AJD, Lightfoot NJ. Local anaesthetic delivery regimens for peripheral nerve catheters: a systematic review and network meta-analysis. Anaesthesia. 2020 Mar;75(3):395-405. doi: 10.1111/anae.14864. Epub 2019 Oct 14. PMID 31612480
- [Background] Jagannathan R, Niesen AD, D'Souza RS, Johnson RL. Intermittent bolus versus continuous infusion techniques for local anesthetic delivery in peripheral and truncal nerve analgesia: the current state of evidence. Reg Anesth Pain Med. 2019 Apr;44(4):447-451. doi: 10.1136/rapm-2018-100082. Epub 2019 Feb 3. PMID 30914472
- [Background] Duan L, Zhang L, Shi CG, Huang LG, Ao H, Wang ZP, Deng Y, Sun ML. Comparison of continuous pericapsular nerve group (PENG) block versus continuous fascia iliaca compartment block on pain management and quadriceps muscle strength after total hip arthroplasty: a prospective, randomized controlled study. BMC Anesthesiol. 2023 Jul 11;23(1):233. doi: 10.1186/s12871-023-02190-1. PMID 37434138
- [Background] Senthil KS, Kumar P, Ramakrishnan L. Comparison of Pericapsular Nerve Group Block versus Fascia Iliaca Compartment Block as Postoperative Pain Management in Hip Fracture Surgeries. Anesth Essays Res. 2021 Oct-Dec;15(4):352-356. doi: 10.4103/aer.aer_119_21. Epub 2022 Mar 1. PMID 35422548
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Butcher NJ, Monsour A, Mew EJ, Chan AW, Moher D, Mayo-Wilson E, Terwee CB, Chee-A-Tow A, Baba A, Gavin F, Grimshaw JM, Kelly LE, Saeed L, Thabane L, Askie L, Smith M, Farid-Kapadia M, Williamson PR, Szatmari P, Tugwell P, Golub RM, Monga S, Vohra S, Marlin S, Ungar WJ, Offringa M. Guidelines for Reporting Outcomes in Trial Protocols: The SPIRIT-Outcomes 2022 Extension. JAMA. 2022 Dec 20;328(23):2345-2356. doi: 10.1001/jama.2022.21243. PMID 36512367